CLINICAL TRIAL: NCT05296460
Title: Efficacy of Dapsone Gel 7.5%in Comparison to Trichloroacetic Acid 20% for Treatment of Acne Vulgaris :Split Face Study
Brief Title: DAPSONE GEL7.5%Versus Trichloroacetic Acid 20% ON ACNE VULGARIS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sahar Ramadan Bestawy, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAPTCA
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dapsone gel and trichloroacetic acid (Experimental): trichloroacetic acid peeling on right side of face and dapsone gel on left side
  Interventions: Drug: Dapsone gel

INTERVENTIONS:
Drug: Dapsone gel — The patients will use topical dapsone gel 7.5% once daily on left side of face ,The patients will use TCA20% peeling as a peeling session every 2 weeks (6 sessions) on right side of face

SUMMARY:
Acne vulgaris, a chronic inﬂammatory skin disorder, is one of the most prevalent diseases that eﬀects more than 80% of the population worldwide . A variety of factors such as genetics, hormones, infections, as well as environmental factors have been identiﬁed as the causes of acne development . Acne usually generates as a result of blockage in the pilosebaceous unit (including hair follicle, hair shaft, and sebaceous gland) due to the over-produced sebum by sebaceous gland, which further triggers the excessive proliferation of the bacterium Propionibacterium acnes (P. Acnes).

DETAILED DESCRIPTION:
Chemical peeling can target the pathogenic factors recognized in acne and treat present primary and secondary lesions, it also improves the pigmentary changes seen with acne, and hastes the time taken to repair skin to normal. Trichloroacetic acid (TCA), salicylic acid (SA), and azelaic acid (AA) have proved efficacy in the treatment of acne as a result of their exfoliative and keratolytic properties .

The mechanism of TCA peel in the treatment of acne vulgaris is due to its ability to diminish corneocyte cohesion and keratinocyte plugging, thus helping in comedolytic action. In addition, application of TCA to the skin causes precipitation of proteins and coagulative necrosis of epidermal cells, leading to removal of damaged skin and its replacement by normal tissue.

Dapsone is a "4,40-diamino diphenyl sulfone" compound and an aniline derivative from synthetic sulphones.. Sulphonamides were first used in humans as antimicrobial agents to treat streptococcal infections. Dapsone derived from sulphonamides was first used in the treatment of leprosy in 1940 . Subsequently, it was used in the treatment of bullous dermatoses, especially dermatitis herpetiformis, and in the treatment of non-infectious inflammatory dermatoses, especially neutrophilic dermatoses . Today, Dapsone treatment is among the treatment options for many dermatological diseases.

Dapsone carries both bacteriostatic and anti-inflammatory properties. Its antimicrobial effect stems from its sulfonamide-like ability to inhibit the synthesis of dihydrofolic acid .

Additionally, dapsone has multiple anti-inflammatory properties. It inhibits the production of reactive oxygen species directly and reversibly inhibits the myeloperoxidase enzyme thus decreasing hypochlorous acid formation.

further more topical dapsone has been used with different concentration in treating acne vulgaris: both dapsone gel 7.5% and dapsone gel 5%has been used and found to be safe and effective

ELIGIBILITY:
Inclusion Criteria:

* Both males and females will be included.
* Patients older than 12 years of age.
* Patients with mild and moderate AV.
* Patients had not received any topical or systemic treatment for AV during the previous 2 weeks

Exclusion Criteria:

* Severe acne.
* Patients under treatment with contraceptive pills or any kind of systemic or topic acne medication (isotretinoin, antibiotics, topical products).
* History of hypertrophic/keloid scar formation.
* Pregnancy, breast feeding.
* Recurrent herpes infection.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the medication:number of inflammatory ,non inflammatory and total lesions. counting the number of inflammatory ,non inflammatory and total lesions at baseline and every 4 weeks during the treatment | 12 weeks
  assessment of tolerability:interviewing the patients about any sign/symptoms of adverse reactions(erythema,peeling,burning sensation,dryness and pruritus)

CONTACTS AND LOCATIONS:
Overall Officials: dalia attallah, pof dr, Study Director — assiut

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Atallah DA, Bestawy SR, Abouelmajd SA, Badran AY. Dapsone 7.5% Gel Versus Trichloroacetic Acid Peels. Dermatol Surg. 2025 Oct 3. doi: 10.1097/DSS.0000000000004896. Online ahead of print. PMID 41042170